CLINICAL TRIAL: NCT00849992
Title: Randomized Prospective Study Comparing 5% Imiquimod and Photodynamic Therapy for Actinic Cheilitis
Brief Title: Treatment Study for Actinic Cheilitis Comparing Imiquimod 5% and Photodynamic Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20115
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Actinic Cheilitis
Keywords: Actinic cheilitis; Imiquimod 5%; Photodynamic therapy
MeSH Terms: conditions — Actinic cheilitis | interventions — Imiquimod; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imiquimod 5% (Other): Patients randomized to this arm will receive treatment with imiquimod 5%
  Interventions: Drug: Imiquimod 5%
- Photodynamic therapy (Other): Patients will be randomized to receive photodynamic therapy twice at a 2 week interval to the affected area.
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Drug: Imiquimod 5% — Imiquimod 5% cream used three days a week for 4 weeks
  Other Names: Aldara
  Arms: Imiquimod 5%
Procedure: Photodynamic therapy — Photodynamic therapy involves applying Metvix cream to the affected area followed by illumination. It will be done twice during the study at a 2 week interval.
  Arms: Photodynamic therapy

SUMMARY:
Actinic cheilitis is a common precancerous lesion of the lip. The purpose of this study is to compare imiquimod 5% therapy and photodynamic therapy. The data will include effect data, histology (skin analysis), epidemiological data and follow-up data.

DETAILED DESCRIPTION:
Randomized study comparing imiquimod 5% with photodynamic therapy for actinic cheilitis. Histological, efficacy, epidemiological and clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Clinical findings of actinic cheilitis.
* Histological findings demonstrating epithelial changes equal to or greater than mild epithelial dysplasia in severity (mild - moderate - severe).
* Age above 18.
* Willingness to take post-treatment biopsy.

Exclusion Criteria:

* Disorders predisposing to photosensitivity (porphyria, SLE).
* Pregnancy or nursing.
* Known allergy to any excipients in the study creams.
* prescribed topical retinoids, 5-fluorouracil, cryodestruction, surgical excision and curettage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
clinical and pathological complete cure rates. | 3 and 12 months after therapy

SECONDARY OUTCOMES:
clinical, safety, epidemiological and histopathological data | post-treatment
  Through collecting patient data and post-treatment biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Stein H Sundstrøm, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway